CLINICAL TRIAL: NCT06879288
Title: Efficacy of Dexmedetomidine Versus Magnesium Sulfate as Adjuvants to Intraperitoneal Bupivacaine for Postoperative Analgesia in Patients Undergoing Elective Laparoscopic Cholecystectomy
Brief Title: Dexmedetomidine Versus Magnesium Sulfate as Adjuvants to Intraperitoneal Bupivacaine for Postoperative Analgesia After Elective Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maha Mahmoud Rabee El Gazzar, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS215/6/23
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Dexmedetomidine; Magnesium Sulfate; Adjuvants; Intraperitoneal Bupivacaine; Postoperative Analgesia; Elective Laparoscopic Cholecystectomy
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine group (Active Comparator): Patients received intraperitoneal bupivacaine only at the end of the operations.
  Interventions: Drug: Bupivacaine
- Dexmedetomidine group (Experimental): Patients received intraperitoneal bupivacaine plus dexmedetomidine at the end of the operations.
  Interventions: Drug: Dexmedetomidine
- Magnesium group (Experimental): Patients received intraperitoneal bupivacaine plus magnesium sulfate at the end of the operations.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Bupivacaine — Patients received intraperitoneal bupivacaine only at the end of the operations.
  Arms: Bupivacaine group
Drug: Dexmedetomidine — Patients received intraperitoneal bupivacaine plus dexmedetomidine at the end of the operations.
  Arms: Dexmedetomidine group
Drug: Magnesium sulfate — Patients received intraperitoneal bupivacaine plus magnesium sulfate at the end of the operations.
  Arms: Magnesium group

SUMMARY:
This study aimed to assess the efficiency of dexmedetomidine against magnesium sulfate as adjuvants to intraperitoneal bupivacaine for postoperative analgesia in individuals having elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Pain after laparoscopy is less intense than after laparotomy, but laparoscopy is not pain free and analgesia after this type of surgery is inadequately studied. Intraperitoneal (IP) instillation/nebulization of local anesthetics has been used as a method for reducing postoperative pain and opioid use following laparoscopy through acting on visceral nociceptors of the peritoneum.

Bupivacaine is indicated for local infiltration, peripheral nerve block, sympathetic nerve block, and epidural and caudal blocks. It is available mixed with a small amount of epinephrine to increase the duration of its action. It typically begins working within 15 minutes and lasts for 2 to 8 hours.

Dexmedetomidine is a selective alpha-2 (α2) adrenergic agonist known to have analgesic and sedative characteristics that can augment the duration of action of local anesthetics.

Magnesium is an N-methyl-D-aspartate receptor antagonist in addition to its effects on calcium influx. The anti-inflammatory and opioid-sparing effects make it a popular component of opioid free anaesthesia. It is extensively used for perioperative analgesia in a dose of 30- to 50-mg/kg intravascular bolus followed by a 10- to 15-mg/kg/h infusion.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) class I-III.
* Scheduled to undergo elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patient refusal.
* Body mass index ≥40.
* Allergy to the study drugs.
* Advanced cardiac, renal and hepatic diseases.
* Patients with peritoneal drain or peritoneal wash after surgery.
* Uncooperative patients.
* Chronic pain medications.
* Hypomagnesaemia or hypermagnesaemia.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Degree of pain was assessed using the numerical rating score (NRS) (from 0 = no pain, to 10 = the most severe pain).NRS was assessed at 1, 2, 4, 8, 16, and 24 hours postoperative.

SECONDARY OUTCOMES:
Time to the first rescue analgesia request | 24 hours postoperatively
  Time to the first rescue analgesia request (time from the end of surgery till first dose of morphine administrated)
Total morphine consumption | 24 hours postoperatively
  If Numerical rating score (NRS)-S >4, IV 3 mg morphine was given as a rescue analgesia.
Level of sedation | 24 hours postoperatively
  Level of sedation using Ramsey scale at 1, 2, 4, 8, 16, and 24 hours postoperative from 1 to 6:
  1. Patient is anxious and agitated.
  2. Patient is co-operative and oriented.
  3. Patient responds to commands only.
  4. Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
  5. Patient exhibits sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response.
Lenght of hospital stay | 1 week postoperatively
  Length of hospital stay was recorded from admission till discharge from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.